CLINICAL TRIAL: NCT02139514
Title: Virtual Reality Social Cognition Training for Adults With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1211011083
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Autism Spectrum Disorders
Keywords: Social Skills; Adults
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills

ARMS (2):
- Virtual Reality Social Cognition Training (Active Comparator): Virtual Reality Social Cognition Training
  Interventions: Behavioral: Virtual Reality Social Cognition Training
- Control (No Intervention): Participants in the Control condition will be offered treatment following the Control condition.

INTERVENTIONS:
Behavioral: Virtual Reality Social Cognition Training — Social skills training via virtual reality with trained therapist.
  Arms: Virtual Reality Social Cognition Training

SUMMARY:
The purpose of this study is to predict and explain on the basis of brain function and structure the behavioral and brain effects of an evidence-based intervention for adults with high-functioning autism, Virtual Reality-Social Cognition Training (Kandalaft et al., 2012; Journal of Autism and Developmental Disorders). Adults with autism will be randomly assigned to receive either (a) two hours per week of intervention services for five weeks, or (b) a treatment as usual control. The intervention will focus on enhancing social skills, social cognition, and social functioning. Outcome measures will evaluate changes in these social skills, cognition, and functioning using standardized assessments. We will perform structural and functional magnetic resonance imaging (MRI) scans at three time points-before, during, and after treatment (i.e., Time Point #1, 2, and 3).

DETAILED DESCRIPTION:
The purpose of this study is to predict and explain on the basis of brain function and structure the behavioral and brain effects of an evidence-based intervention for adults with high-functioning autism, Virtual Reality-Social Cognition Training (Kandalaft et al., 2012; Journal of Autism and Developmental Disorders). Adults with autism will be randomly assigned to receive either (a) two hours per week of intervention services for five weeks, or (b) a treatment as usual control. The intervention will focus on enhancing social skills, social cognition, and social functioning. Outcome measures will evaluate changes in these social skills, cognition, and functioning using standardized assessments. We will perform structural and functional magnetic resonance imaging (MRI) scans at three time points-before the treatment, after the treatment, and a 3-month follow-up (i.e., Time Point #1, 2, and 3).

All the recruitment will be taking place at Yale Child Study Center (YCSC), while the intervention will be delivered online by therapists located at the Center for BrainHealth at the University of Texas at Dallas (UTD). The intervention is called Virtual Reality-Social Cognition Training (VR-SCT) and has been approved by the IRB at UTD (approval number #06-54).

ELIGIBILITY:
Inclusion Criteria:

1. Adults:

   1. Age: 18-40, inclusive
   2. A male or female outpatient
2. High-functioning (so that the treatment can effectively benefit the subjects):

   1. Full Scale Intelligence Quotient (IQ) of WASI at least 80
   2. Able to give informed consent prior to initiation of any protocol required procedures
3. Autism Spectrum Disorder:

   1. Having a current primary diagnosis of Autism Spectrum Disorder (including Asperger's Disorder) from a licensed psychologist/psychiatrist or from a school diagnostician, as defined by the DSM-IV criteria.
   2. For this project, diagnosis will not be determined by our assessment. The participants we enroll will already carry a current primary diagnosis of Autism Spectrum Disorder. This verification of their diagnosis may also come from study personnel who have seen and/or treated the patient prior to his or her involvement in the project and can verbally confirm that they carry the proper diagnosis.
4. Mean Length of Utterance (MLU) must be at least 4-5 words (the intervention method requires this)

Exclusion Criteria:

1. Speech-language criteria:

   1. Those who are not fluent in written and oral English will not be eligible to participate, as many of the instruments are not validated in other languages.
   2. Significant hearing loss or other severe sensory impairment
   3. Inability to read self-report instruments
2. Health criteria:

   1. Those whose clinical status (e.g., serious suicidal or homicidal risk) requires inpatient or day hospital treatment
   2. Those with a history of seizures, or current use of anticonvulsants
   3. A fragile health status
   4. A history of significant head trauma or serious brain or psychiatric illness
   5. Having any other current psychiatric condition or complications, such as

   i. Diagnosed with substance dependence within the last three months. ii. Current use of prescription medications that may affect cognitive processes under study.

   iii. Current primary diagnosis of bipolar disorder I or II iv. Axis I psychopathology v. Depression
3. Any metal or electromagnetic implants, including:

   1. Cardiac pacemaker
   2. Defibrillator
   3. Artificial heart valve
   4. Aneurysm clip
   5. Cochlear implants
   6. Shrapnel
   7. Neurostimulators
   8. History of metal fragments in eyes or skin

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
functional magnetic resonance imaging (MRI) | up to 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States